CLINICAL TRIAL: NCT02920658
Title: Nonaromatic Naphthalan - Composition Study and Biological Effects on Epithelial Tissues
Brief Title: Topical "Non-Aromatic Very Rich in Steranes" (NAVS) Naphthalan for the Treatment of Oral Mucosal Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ivan Alajbeg (Other)
Collaborators: Ministry of Science, Education and Sport, Republic of Croatia (Other Government)
Responsible Party: Sponsor-Investigator, Ivan Alajbeg, Professor of Oral Medcine, University of Zagreb
Organization: University of Zagreb (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 065-0650445-1277
Record Dates: First submitted 2016-06-08; First posted 2016-09-30 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Oral Lichen Planus; Recurrent Aphthous Stomatitis
Keywords: NAVS Naphthalan; Betamethasone dipropionate; Topical treatment
MeSH Terms: conditions — Lichen Planus, Oral; Stomatitis, Aphthous | interventions — betamethasone-17,21-dipropionate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NAVS Naphthalan (Experimental): NAVS oil in adhesive powder in a volume ratio 2:1, to apply on the affected mucosa three times daily during 4 weeks for OLP patients; NAVS oil in adhesive powder in a volume ratio 2:1, to apply on the affected mucosa three times daily during 5 days for RAS patients
  Interventions: Drug: NAVS Naphthalan
- 0.05% Betamethasone dipropionate (Active Comparator): 0.05% Betamethasone dipropionate in adhesive powder in a volume ratio 1:1, to apply on the affected mucosa three times daily during 4 weeks for OLP patients; 0.05% Betamethasone dipropionate in adhesive powder in a volume ratio 1:1, to apply on the affected mucosa three times daily during 5 days for RAS patients
  Interventions: Drug: 0.05% Betamethasone dipropionate

INTERVENTIONS:
Drug: NAVS Naphthalan
  Arms: NAVS Naphthalan
Drug: 0.05% Betamethasone dipropionate
  Other Names: Beloderm
  Arms: 0.05% Betamethasone dipropionate

SUMMARY:
This study evaluates the effectiveness of topical NAVS naphthalan in the treatment of oral lichen planus (OLP) and recurrent aphthous stomatitis (RAS). Half of participants with OLP and RAS will receive topical NAVS naphthalan in adhesive paste, while the other half will receive 0.05%-betamethasone dipropionate in adhesive paste. Our hypothesis is that NAVS could be efficient in the treatment of OLP and RAS, with effects comparable to that of topical steroids.

DETAILED DESCRIPTION:
Non-Aromatic-Very rich in Steranes (NAVS) naphthalan is a transparent, earth mineral oil prepared by a complex set of procedures of separations and refining, starting with a special oil that is used as the raw material for brown naphthalane, which has been successfully used in the treatment of psoriasis. In order to remove potentially mutagenic polycyclic aromatic hydrocarbons (PAHs), liquid chromatography was used. UV / VIS (ultra violet / visible light) spectrophotometry confirmed that PAHs were bellow detection threshold. Additionally, the precise distillation process has concentrated steranes, which are important bioactive constituents. Since steranes contain similar chemical structure as well-known bioactive substances, such as vitamin D3 and steroid hormones, the assumption is that NAVS is effective in the treatment of oral diseases which have immune genesis such as OLP and RAS.

Today, topical steroid preparations are considered as first-line therapy for many chronic immune-mediated inflammatory diseases of the oral mucosa. Risks of short-term use of topical corticosteroids are clinically insignificant, while their long-term use is not recommended because of potential side effects, such as mucosal atrophy, secondary infection with Candida albicans, possible systemic absorption and suppression of the adrenal gland.

Study participants are adult patients of the Department of Oral Medicine, School of Dental Medicine in Zagreb, with a clinically and histologically proven OLP or RAS in the acute stage of the disease.The treatment outcome of the OLP patients will be measured by clinical improvement and subjective symptomatic relief. The outcome of RAS patients treated by NAVS naphthalan or by betamethasone will be measured clinically by the decrease in number and size of lesions as well as by subjective symptomatic relief over treatment period. One member of the team, who will not evaluate the therapeutic effect, will took care of the allocation of test and control preparations. At the end of the study, a randomization code will be opened and statistically analysed. In both clinical and subjective domains, of both clinical conditions, the improvement rate will be measured by comparing these readings, as the percentual reduction of clinical scores and symptoms. Since the data will not be normally distributed, methods of nonparametric statistics will be used: Wilcoxon test for dependent and Mann-Withney test for independent samples. Baseline intergroup differences will be assessed by Mann-Withney test. For the interpretation of the average values, medians and interquartile ranges (IQR) will be used. Fisher exact test will be used to compare gender representation among the groups. Statistical analysis will be performed using MedCalc Software 13.0.0.0 (Acacialaan 22, 8400 Ostend, Belgium). P value lower then 0.05 (p< 0.05) will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* for OLP patients: adult patients with a clinically and histologically proven OLP (Al-Hashimi et al, 2007)
* for RAS patients: in the acute stage of the disease, according to Lehner (1968), at least 2 episodes per year

Exclusion Criteria:

* for OLP patients: younger than 18 years, hepatobiliary system diseases, lichenoid reaction (amalgam, drugs) or lichen planus with lesions in contact to restorative materials (Zakrzewska et al, 2005), the current comparative systemic or local anti-inflammatory treatment (antibiotics, corticosteroids, non-steroidal antirheumatic drugs, chemotherapeutics) (Lo Muzio et al, 2001; Nolan et al, 2006; Rodriguez et al, 2007) and pregnancy.
* for RAS patients: patients younger than 18 years, haematological deficits (assessed by complete blood count (CBC), iron (Fe), vitamin B12, hypersensitivity to toothpaste and oral mouth rinse solutions (assessed by medical history) (Nolan et al, 2006), pregnancy, inflammatory bowel disease (assessed by medical history), significant immunodeficiencies, current comparative systemic or topical anti-inflammatory treatment (antibiotics, corticosteroids, nonsteroidal antirheumatics, chemotherapeutics) (Lo Muzio et al, 2001; Nolan et al, 2006; Rodriguez et al, 2007).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The change of presence of reticulation, erythema and ulceration on mucosal surfaces | 28 days per patient
  Clinical improvement of OLP lesions after treatment will be scored (Pibooniyom et al.,2005). This clinical scale measures the presence of reticular, erythematous and ulcerative lesions on oral mucosal surfaces, providing a score by adding those values.
  Investigator will assess patients' lesions on oral mucosal surfaces, on day 0 and day 28 and provide score for each assessment. The change of this score between the two time points is a measure of clinical efficacy of applied treatment modality.
  Calibration process : three examiners independently reviewed and evaluated photo of the individual patient. The second evaluation of photographs was a week after to assess the objectivity of the reading on the first visit. Once the examiners reviewed the photographs twice with one-week gap, the obtained results were analysed using Spearman "rank" correlation to determine intra- and inter-observer reliability.
The change in the number of RAS lesions | 5 days per patient
  The number of RAS lesions will be recorded on day 0 and on day 5 after the start of treatment (Khandwala et al, 1997). The change in the number of lesions between the two time points is a measure of clinical efficacy of applied treatment modality.
The change in the diameter of RAS lesions | 5 days per patient
  The change in the diameter of RAS lesions (in millimeters) will be recorded on day 0 and on day 5 after the start of treatment (Khandwala et al, 1997). The change in the cumulative diameter of lesions between the two time points is a measure of clinical efficacy of applied treatment modality.
The change of pain intensity and discomfort in OLP patients | 28 days per patient
  The intensity of pain and discomfort will be determined using a 100 mm visual analog scale (VAS) on day 0 and day 28. The change in the amount between the two time points is a measure of clinical efficacy of applied treatment modality.
The quality of life change in OLP patients | 28 days per patient
  The quality of life for OLP patients will be determined using "Oral health impact profile"(OHIP-14) questionnaire on day 0 and day 28. The change in the amount between the two time points is a measure of clinical efficacy of applied treatment modality.
The change of pain intensity and discomfort in RAS patients | 5 days per patient
  The intensity of pain and discomfort will be determined using a 100 mm visual analog scale (VAS) 30 and 60 minutes after the application of the therapeutic agent at home. The change in the amount between the two time points is a measure of clinical efficacy of applied treatment modality.
The quality of life change in RAS patients | 5 days per patient
  The quality of life for RAS patients will be determined using "Oral health impact profile"(OHIP-14) questionnaire on day 0 and day 5. The change in the amount between the two time points is a measure of clinical efficacy of applied treatment modality.

SECONDARY OUTCOMES:
Adverse reactions to treatment modalities in OLP patients | 28 days per patient
  In OLP patients application of both treatment modalities lasts for 28 days. The occurrence of oral Candidal infection or irritation will be recorded by clinician on day 28. The frequency of each will be compared between two treatment groups.

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Alajbeg, PhD, Principal Investigator — University of Zagreb
Locations (1):
- School of Dental medicine, University of Zagreb, Zagreb, City of Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Yes, de-identified data are available upon request.

REFERENCES:
- [Background] Al-Hashimi I, Schifter M, Lockhart PB, Wray D, Brennan M, Migliorati CA, Axell T, Bruce AJ, Carpenter W, Eisenberg E, Epstein JB, Holmstrup P, Jontell M, Lozada-Nur F, Nair R, Silverman B, Thongprasom K, Thornhill M, Warnakulasuriya S, van der Waal I. Oral lichen planus and oral lichenoid lesions: diagnostic and therapeutic considerations. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Mar;103 Suppl:S25.e1-12. doi: 10.1016/j.tripleo.2006.11.001. Epub 2007 Jan 29. PMID 17261375
- [Background] Khandwala A, Van Inwegen RG, Alfano MC. 5% amlexanox oral paste, a new treatment for recurrent minor aphthous ulcers: I. Clinical demonstration of acceleration of healing and resolution of pain. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1997 Feb;83(2):222-30. doi: 10.1016/s1079-2104(97)90009-3. PMID 9117754
- [Background] Lehner T. Autoimmunity in oral diseases, with special reference to recurrent oral ulceration. Proc R Soc Med. 1968 May;61(5):515-24. doi: 10.1177/003591576806100543. No abstract available. PMID 4297643
- [Background] Lo Muzio L, della Valle A, Mignogna MD, Pannone G, Bucci P, Bucci E, Sciubba J. The treatment of oral aphthous ulceration or erosive lichen planus with topical clobetasol propionate in three preparations: a clinical and pilot study on 54 patients. J Oral Pathol Med. 2001 Nov;30(10):611-7. doi: 10.1034/j.1600-0714.2001.301006.x. PMID 11722711
- [Background] Neppelberg E, Johannessen AC, Jonsson R. Apoptosis in oral lichen planus. Eur J Oral Sci. 2001 Oct;109(5):361-4. doi: 10.1034/j.1600-0722.2001.00081.x. PMID 11695759
- [Background] Nolan A, Baillie C, Badminton J, Rudralingham M, Seymour RA. The efficacy of topical hyaluronic acid in the management of recurrent aphthous ulceration. J Oral Pathol Med. 2006 Sep;35(8):461-5. doi: 10.1111/j.1600-0714.2006.00433.x. PMID 16918596
- [Background] Piboonniyom SO, Treister N, Pitiphat W, Woo SB. Scoring system for monitoring oral lichenoid lesions: a preliminary study. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2005 Jun;99(6):696-703. doi: 10.1016/j.tripleo.2004.07.013. PMID 15897856
- [Background] Rodriguez M, Rubio JA, Sanchez R. Effectiveness of two oral pastes for the treatment of recurrent aphthous stomatitis. Oral Dis. 2007 Sep;13(5):490-4. doi: 10.1111/j.1601-0825.2006.01327.x. PMID 17714352
- [Background] Zakrzewska JM, Chan ES, Thornhill MH. A systematic review of placebo-controlled randomized clinical trials of treatments used in oral lichen planus. Br J Dermatol. 2005 Aug;153(2):336-41. doi: 10.1111/j.1365-2133.2005.06493.x. PMID 16086745
- [Derived] Rogulj AA, Z Alajbeg I, Brailo V, Skrinjar I, Zuzul I, Vucicevic-Boras V, Alajbeg I. Topical NAVS naphthalan for the treatment of oral lichen planus and recurrent aphthous stomatitis: A double blind, randomized, parallel group study. PLoS One. 2021 Apr 8;16(4):e0249862. doi: 10.1371/journal.pone.0249862. eCollection 2021. PMID 33831097